CLINICAL TRIAL: NCT00597792
Title: Registry Study of the NDO Surgical Plicator for the Treatment of GERD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsoring company ceased business operations
Sponsor: NDO Surgical, Inc. (Industry)
Responsible Party: Bruce Gaumond/Associate Director, Clinical Affairs, NDO Surgical, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135-01762
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: GERD
Keywords: Gastroesophageal Reflux Disease (GERD); Plicator; Full-thickness Plication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): Active Plicator Treatment
  Interventions: Device: NDO Full-thickness Plicator

INTERVENTIONS:
Device: NDO Full-thickness Plicator — A low-profile (≤6mm) gastroscope was advanced and an EGD followed by Savary wire placement was performed. The gastroscope was then removed and the Plicator was advanced directly over the wire and into the stomach. The gastroscope was re-introduced through the Plicator, and the Plicator was retroflexed under direct endoscopic visualization to the anterior gastric cardia, approximately 1cm below the gastroesophageal (GE) junction. The Plicator arms were opened and the endoscopic tissue retractor was advanced deeply into the gastric cardia. The gastric wall was then retracted into the open arms of the Plicator. The arms were closed and a single, transmural pledgeted suture was deployed. The Plicator and gastroscope were then removed and the gastroscope re-inserted to evaluate the post-plication GE junction.

SUMMARY:
The purpose of this study is to collect post-marketing data on patient outcomes and satisfaction following treatment with the Plicator™. The outcomes will be tracked through analysis of patient Quality of Life (QoL) questionnaires and medication use. The QoL and medication use questionaires will be administered and documented twice before the procedure and then again at outlined intervals following the procedure. Additionally, financial measures will be evaluated (i.e. pre-procedural and procedural time and costs, staffing/personnel needs during procedure, anesthesia and related costs, recovery time and associated cost, etc.) and post-procedure GERD-related medical history questionnaires will be completed.

This post-market evaluation is a multi-center study design using the NDO Surgical, Inc. Plicator as the treatment device. Treatment efficacy will be evaluated by comparing QoL and medication use before and after treatment with the device. Patient follow-ups will be completed at 1 week and at 6, 12, 24, 36, 48 and 60 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is suitable for surgery (American Society of Anesthesiologists Physical Status Classification I or II).
* Subject agrees to study participation and signs/dates an informed consent form.

Exclusion Criteria:

* Significant esophageal dysmotility as determined by manometry
* Esophagitis grade III or IV (Savary-Miller)
* Barrett's epithelium
* Hiatus hernia > 2cm
* Persistent dysphagia, weight loss, esophageal bleeding, vomiting, gas or bloating
* Esophageal or gastric varices
* Previous endoscopic or surgical anti-reflux procedure
* Other esophageal or gastric surgery
* Chronic use of anticoagulant or platelet anti-aggregation therapy (other than for cardiac prophylaxis); and
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6, 12, 24, 36, 48, 60 months post-treatment

SECONDARY OUTCOMES:
GERD Medication Use | 6, 12, 24, 36, 48, 60 months post-treatment
Economic outcomes (e.g. procedure time/costs, staffing needs, anesthesia costs, recovery time/costs) | 6, 12, 24, 36, 48, 60 months post-procedure
Subject satisfaction | 6, 12, 24, 36, 48, 60 months post-treatment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Medical Center of Central Georgia, Macon, Georgia
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Northside Gastroenterology, Inc., Indianapolis, Indiana
  - Lenox Hill Hospital, New York, New York
  - Stony brook University Medical Center, Stony Brook, New York
  - Nashville Medical Research and the Maria Nathanson Center of Excellence, Nashville, Tennessee
  - Digestive Associates of Houston, Houston, Texas